CLINICAL TRIAL: NCT03693846
Title: A Phase II Study of Nivolumab and Ipilimumab in Mucinous Colorectal and Appendiceal Tumors
Brief Title: Nivolumab and Ipilimumab in Mucinous Colorectal and Appendiceal Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow enrollment and lack of efficacy
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 28218
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and Ipilimumab (Experimental): Treatment will consist of Nivolumab 480mg every 4 weeks and Ipilimumab 1mg/kg every 8 weeks. Subjects will continue on study therapy until disease progression, unacceptable toxicity, withdrawal of consent, or 24 months of therapy.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — IV infusion per institutional guidelines and the Package Insert
  Other Names: Opdivo
Drug: Ipilimumab — IV infusion per institutional guidelines and the Package Insert
  Other Names: Yervoy

SUMMARY:
This is a single-arm phase II study of twenty-one subjects with mucinous adenocarcinoma of the colon, rectum, or appendix with prior systemic therapy with a fluoropyrimidine, oxaliplatin, and irinotecan. Treatment will consist of nivolumab 480mg every 4 weeks and ipilimumab 1mg/kg every 8 weeks until disease progression, unacceptable toxicity, or 2 years of therapy.

DETAILED DESCRIPTION:
Treatment will consist of nivolumab 480mg every 4 weeks and ipilimumab 1mg/kg every 8 weeks (within a 56-day cycle, (Nivolumab administered on days 1 and 29, and Ipilimumab administered on day 1 of each cycle). Imaging assessments will be conducted every 8 weeks (+/-2 weeks) for the first 24 weeks then every 8-12 weeks (+/-2 weeks). If progression is noted on imaging in the setting of clinical stability, subjects may remain on study and have confirmatory imaging in 4-8 weeks per iRECIST criteria

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated an IRB-approved written informed consent form prior to the performance of any protocol-related procedures that are not part of standard care.
* Colorectal or appendiceal mucinous adenocarcinoma with peritoneal-only metastatic disease. It is recognized that in some patients, peritoneal disease will predominate without distinction of the site of origin, and such patients will be eligible.
* Microsatellite stable by PCR and/or mismatch repair proficient by immunohistochemistry
* ECOG performance status of 0 or 1
* Prior therapy with a fluoropyrimidine, oxaliplatin, and irinotecan unless contraindicated or refused. Prior treatment with antiangiogenic and/or anti-EGFR antibody therapy is permitted but not required
* Measurable disease by RECIST v. 1.1
* Laboratory parameters:

  * Absolute neutrophil count > 1500/μL
  * Platelets > 100,000/μL
  * Hemoglobin > 9.0 g/dL
  * PT/INR or PTT < 1.5xULN
  * Creatinine < 1.5xULN OR creatinine clearance > 50 mL/min by Cockcroft-Gault formula
  * Total bilirubin < 1.5xULN
  * Subjects with Gilbert's Syndrome must have a total bilirubin level of < 3.0xULN
  * Albumin > 3.0 g/dL
  * AST and/or ALT: < 3.0×ULN
* Subjects with HIV are permitted provided they meet the following criteria:

  * CD4+ cell count > 250 cells/mm3
  * No history of AIDS-defining conditions other than low CD4+ count
  * If subject is on antiretroviral therapy, there must not be expected significant drug-drug interactions with study treatment

Exclusion Criteria:

* Bowel obstruction within the past 60 days
* Subjects who are currently pregnant, planning to become pregnant, or breast-feeding.

  * Females participants of child-bearing potential are required to use an effective contraception method or abstain from intercourse during treatment and for at least 5 months following the last dose
  * Males participants with partners of child-bearing potential are required to use an effective contraception method or abstain from intercourse during treatment and for at least 7 months following the last dose
* Subjects who, in the opinion of the physician, would not be clinically appropriate for receipt of the therapy regimen associated with participation
* Subjects with contraindications to immune checkpoint therapy, as follows:

  * Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity
  * Prior organ allograft or allogeneic bone marrow transplantation
  * Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
  * Active autoimmune disease, except for vitiligo, type 1 diabetes mellitus, asthma, atopic dermatitis, or endocrinopathies manageable by hormone replacement; other autoimmune conditions may be allowable at the discretion of the principal investigator
  * Condition requiring systemic treatment with corticosteroids

    * Systemic steroids at physiologic doses (equivalent to dose of oral prednisone 10 mg) are permitted.
    * Intranasal, inhaled, topical, intra-articular, and ocular corticosteroids with minimal systemic absorption are permitted.
* Established non-peritoneal metastatic disease, including but not limited to metastases to the liver, lung, brain, extra-abdominal lymph nodes, and bone
* A second primary malignancy that, in the judgment of the investigator, may affect interpretation of results
* Prior treatment with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody
* Toxicities attributed to prior anti-cancer therapy other than alopecia, fatigue, and peripheral neuropathy must have resolved to Grade 1 or baseline before administration of study drug. In addition, a washout period will be required for prior therapies as specified:

  * No chemotherapy within 14 days prior to first dose
  * No investigational product(s) (IPs) and/or biologic therapy within 28 days or 5 half-lives, whichever is longer, prior to first dose
  * No major surgery within 28 days prior to first dose. Any surgery-related AE(s) must have resolved at least 14 days prior to first dose.
  * No radiation therapy with curative intent within 28 days prior to first dose. Prior focal palliative radiotherapy must have been completed at least 14 days prior to first dose.
* Active hepatitis B or hepatitis C, defined as the following:

  * Hepatitis B surface antigen positive or HBV DNA PCR >100 IU/mL
  * Hepatitis C antibody positive unless HCV RNA PCR is negative (i.e. undetectable viral load)
* Prisoners or participants who are involuntarily incarcerated. (Note: under specific circumstances a person who has been imprisoned may be included as a participant. Strict conditions apply and BMS approval is required.)
* Participants who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Karasic, MD, Principal Investigator — Abramson Cancer Center
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven subjects were consented/enrolled and active on study treatment for at least one cycle.
Groups:
- Nivolumab and Ipilimumab: Treatment will consist of nivolumab 480mg every 4 weeks and ipilimumab 1mg/kg every 8 weeks.
  Nivolumab: IV infusion per institutional guidelines and the Package Insert
  Ipilimumab: IV infusion per institutional guidelines and the Package Insert
Period: Overall Study
Arm/Group | Nivolumab and Ipilimumab
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-Free Survival at 6 Months
Description: To determine six-month progression-free survival by iRECIST from start of study treatment until 6 months
Time Frame: Start of treatment until 6 months later
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 11
Participants | 0

2. Secondary Outcome: Progression-Free Survival
Description: to determine Progression-Free survival from start of study treatment until time of documented disease progression or death assessed up to 2 years
Time Frame: start of treatment until disease progression or death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 11
months | 1.91 [0.72 to 2.99]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the duration of time from start of treatment to death
Time Frame: From start of treatment until death assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 11
Months | 3.45 [1.61 to 4.04]

4. Secondary Outcome: Objective Response Rate
Description: The objective response rate is determined by the percentage of individuals on study attaining a complete or partial response as noted by by iRECIST and RECIST v1.1 Criteria
Time Frame: From start of treatment until progression or death assessed up to 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 11
Percentage of participants | 0

5. Secondary Outcome: Duration of Response
Description: Time from the first recorded partial or complete response using RECIST v.1.1 criteria until disease progression or death
Time Frame: From the first recorded partial or complete response until progressive disease or death, whichever came first, assessed up to 2 years
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Nivolumab and Ipilimumab
Number analyzed (Participants) | 11
Months | NA [NA to NA] — The duration of response was not reportable as there were no objective responses

ADVERSE EVENTS:
Time Frame: From ICF signature to 100 days following the last administration of study treatment.
Description: All Serious Adverse Events or pregnancies that occur following the subject's written consent to participate in the study through 100 days of discontinuation of dosing must be reported.
  At each contact with the subject, the investigator must seek information on adverse events by specific questioning and, as appropriate, by examination.
Arm/Group | Nivolumab and Ipilimumab
All-Cause Mortality (participants affected / at risk) | 5/11
Serious Adverse Events (participants affected / at risk) | 9/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and Ipilimumab (N=11)
Small Intestine Obstruction (Gastrointestinal disorders) | 2 (2)
Small Intestine Perforation (Gastrointestinal disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (3)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and Ipilimumab (N=11)
Nausea (Gastrointestinal disorders) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 6 (6)
Ascites (Gastrointestinal disorders) | 4 (4)
Abdominal Bloating (Gastrointestinal disorders) | 3 (3)
Thromboembolic Event (Vascular disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Investigations) | 3 (3)
Hyponatremia (Investigations) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator shall provide sponsor with a copy of each publication at the earliest practicable time, but in any event not less than thirty (30) days prior to its submission to a journal, publisher, or meeting or fifteen (15) days prior to any public disclosure of any manuscript or other public disclosure (e.g., presentation).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT03693846/Prot_SAP_001.pdf